CLINICAL TRIAL: NCT01339962
Title: Retrospective Analysis Of Progression Free Survival And Overall Survival In A National Cohort Of Patients With Metastatic Renal Cell Carcinoma Treated In Denmark From 2006-2010. DARENCA Study 2.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Copenhagen University Hospital at Herlev (Other); Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Odense University Hospital (Other); Danish Renal Cancer Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: A6181203; DARENCA STUDY 2
Record Dates: First submitted 2011-04-15; First posted 2011-04-21 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-Interventional Study: Outcomes Research Study
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional (retrospective chart reviews)

SUMMARY:
Non-interventional study. Data obtained by patient chart reviews.

Retrospective analysis of progression free survival, time to treatment failure and overall survival in a national cohort of patients with metastatic renal cell carcinoma treated in Denmark from 2006-2010 Safety, prognostic factors, predictive factors and co-morbidity assessed by Charlson Comorbidity Index.

The following drugs will be evaluated: Sunitinib, Sorafenib, Temsirolimus, Everolimus, Aldesleukin, Interferon-alfa-2b.

DETAILED DESCRIPTION:
No sampling. All eligible patients will be included.

ELIGIBILITY:
Inclusion Criteria:

Metastatic renal cell carcinoma

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Danish patients diagnosed with metastatic renal cell carcinoma referred to the involved centers.
Sampling Method: Non-Probability Sample
Enrollment: 1073 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Overall survival from initiation of first systemic anticancer therapy | 8 months
Progression free survival from initiation of each systemic anticancer therapy separately | 8 months
Time to treatment failure from initiation of each systemic anticancer therapy separately | 8 months

SECONDARY OUTCOMES:
Prognostic factors at baseline associated with efficacy (PFS) of each systemic anticancer therapy and overall survival | 8 months
Serious Adverse Events: Defined as AEs leading to dose adjustment, treatment interruption/ cessation or death. | 8 months
Predictive factors | 8 months
Co-morbidity assessed by Charlson Comorbidity Index | 8 months
Combined PFS and OS on sequential treatment | 8 months
Assessment of first line immunotherapy´s effect on second line targeted therapy | 8 months
Assessment of prognostic factors and overall survival for patients not receiving systemic therapy | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- University of Copenhagen Herlev Hospital, Herlev, Denmark

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181203&StudyName=Retrospective%20Analysis%20Of%20Progression%20Free%20Survival%20And%20Overall%20Survival%20In%20A%20National%20Cohort%20Of%20Patients%20With%20Metastatic%20Renal%20Cell%20Car